CLINICAL TRIAL: NCT02680717
Title: Comparative Effectiveness Trial of Topical Calcipotriene, Clobetasol, and Tacrolimus in the Treatment of Pediatric Plaque Morphea
Brief Title: Comparative Effectiveness Trial in the Treatment of Pediatric Plaque Morphea
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to obtain IRB approval at all sites
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Mayo Clinic (Other); Seattle Children's Hospital (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 730382-2
Record Dates: First submitted 2016-02-09; First posted 2016-02-11 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Clobetasol; calcipotriene; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment 1 (Active Comparator): Calcipotriene 0.005% ointment
  Interventions: Drug: Calcipotriene
- Treatment 2 (Active Comparator): Clobetasol 0.05% ointment
  Interventions: Drug: Clobetasol
- Treatment 3 (Active Comparator): Tacrolimus 0.1% ointment
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Clobetasol — ointment, twice daily (alternating weeks)
  Arms: Treatment 2
Drug: Calcipotriene — ointment, twice daily
  Arms: Treatment 1
Drug: Tacrolimus — ointment, 0.1%, twice daily
  Arms: Treatment 3

SUMMARY:
This is a study designed to evaluate the comparative effectiveness of topical medications for the treatment of circumscribed morphea.

DETAILED DESCRIPTION:
Morphea, also known as localized scleroderma, is a rare autoimmune fibrosing disorder that affects children and adults. Morphea causes significant morbidity through atrophy and fibrosis of the skin and underlying structures. Treatment can halt the progression of disease but cannot reverse disease damage, leaving children with disfiguring scars and sometimes functional impairment. Consequently, it is of extreme importance to intervene early in the disease course with effective therapies to limit morbidity.

Circumscribed morphea is the second most common subtype in children, comprising approximately 1/3 of pediatric morphea cases. It is a disfiguring disease that can cause pain and pruritus. There are no FDA-approved treatments and no consensus exists on the ideal therapy for circumscribed morphea, either in adults or children. Most physicians use topical medications for circumscribed morphea yet there is little evidence to support these therapies. Topical immune modulators such as tacrolimus, imiquimod, and calcipotriene have been investigated in small studies, though these trials were limited by very small sample sizes of 9-19 patients and lack of a control in most. Surveys have demonstrated that topical steroids are the most commonly prescribed medication, even though the only evidence to support their use comes from case reports. With insufficient evidence regarding topical therapies, providers have no guidance when making treatment decisions, practice patterns vary widely even amongst pediatric dermatologists, and children continue with preventable scars.

The investigators specific aim is to identify effective topical therapy for circumscribed morphea. The investigators will utilize a comparative cohort study design to evaluate the comparative effectiveness of three topical medications: clobetasol ointment, calcipotriene ointment, and tacrolimus 0.1% ointment. The investigators will enroll subjects at CHW and other institutions to achieve the study enrollment necessary to power this study.

ELIGIBILITY:
Inclusion Criteria:

* presence of at least 1 active lesion of morphea on the neck, trunk, or extremities with no prior treatment to that lesion for at least 4 weeks

Exclusion Criteria:

* children receiving phototherapy or systemic therapy for their morphea
* children with linear or generalized morphea
* lesions on the face
* greater than 3% body surface area involvement
* open or ulcerated skin within morphea lesions

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 2 months
  This is a 100 mm scale with 3 anchors; each 5 mm of the scale is equivalent to 10% change.
Visual Analog Scale | 4 months
  This is a 100 mm scale with 3 anchors; each 5 mm of the scale is equivalent to 10% change.

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Chiu, MD, Principal Investigator — Medical College of Wisconsin